CLINICAL TRIAL: NCT03911687
Title: Communicating Narrative Concerns Entered by RNs (CONCERN) Clinical Decision Support (CDS) System
Brief Title: (CONCERN) Clinical Decision Support (CDS) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sarah Collins Rossetti, Assistant Professor of Biomedical Informatics and Nursing, Columbia University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAR1389; R01NR016941 (NIH)
Record Dates: First submitted 2019-02-28; First posted 2019-04-11 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Hospital Acquired Condition
Keywords: Early warning system; Clinical decision support; Predictive analysis; Failure to rescue; Inter-professional situational awareness; Nursing surveillance; Healthcare process models of clinical concern (HPM-CC)
MeSH Terms: conditions — Iatrogenic Disease | interventions — Compact Disks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control data will be collected in the CONCERN CDS system that will be "live" in the EHR, but in silent release mode (e.g., not providing notification to clinicians).
- Intervention Group (Experimental): Experimental data will be collected in the CONCERN CDS system that will be "live" in the EHR in "active" release mode (e.g., providing CONCERN CDS system notification to clinicians).
  Interventions: Behavioral: CONCERN CDS system notification

INTERVENTIONS:
Behavioral: CONCERN CDS system notification — The CONCERN CDS will trigger based on analytics of nursing documentation that indicates recognition and concern of patient changes. The CONCERN CDS will alert the care team of the patients "risky state" to increase team-based situational awareness (i.e., shared understanding of the patient situation) of patients predicted to be at risk for patient decompensating in need of rapid intervention to prevent mortality and associated harm.
  Version 1: Burn in phase to evaluate adoption and adaptation to the algorithm being studied. Expected time frame - 3 months
  Version 2: Version 2 refined based on continuous monitoring of data. Expected time frame - 3 months
  Version 3: Version 3 refined based on continuous monitoring of data. Expected time frame - 3 months
  Other Names: CONCERN SMARTapp notification; CONCERN Clinical Decision Support (CDS) system notification
  Arms: Intervention Group

SUMMARY:
There are patients who die or have a bad outcome in the hospital and this could be prevented. Data in the nurses' notes could be used by computers to tell the rest of the care team that a patient is not doing well and that they should act more quickly. This project will build and evaluate a computer system that makes it easier for the care team to see and understand that data and act quickly to save patients. The aims of this study is to answer the questions, what is the level of provider use of the CONCERN CDS notification system (called CONCERN SMARTapp) and resulting impact on selected patient outcomes? Specifically, the study has 1) validated desired thresholds for the CONCERN CDS system and 2) integrated the CONCERN CDS system for early warning of risky patient states within CDS tools.

In this portion of the study (aim 3), the investigator will implement and evaluate the CONCERN CDS system on primary outcomes of in-hospital mortality and length of stay and secondary outcomes of cardiac arrest, unanticipated transfers to the intensive care unit, and 30-day hospital readmission rates.

DETAILED DESCRIPTION:
Annually, more than 200,000 patients die in U.S. hospitals from cardiac arrest and over 130,000 patients inpatients deaths are attributed to sepsis. These deaths are preventable if patients who are at risk are detected earlier. Prior work found that nursing documentation within electronic health records (EHRs) contains information that could contribute to early detection and treatment, but these data are not being analyzed and exposed by EHRs to clinicians to initiate interventions quickly enough to save patients. A new source of predictive data is defined by analyzing the frequency and types of nursing documentation that indicated nurses' increased surveillance and level of concern for a patient. These data documented in the 48 hours preceding a cardiac arrest and hospital mortality were predictive of the event. While clinicians strive to provide the best care, there is a systematic problem within hospital settings of non-optimal communication between nurses and doctors leading to delays in care for patient at risk. Well-designed and tested EHRs are able to trend data and support communication and decision making, but too often fall short of these goals and actually increase clinician cognitive load through fragmented information displays, "note bloat", and information overload. Substitutable Medical Applications & Reusable Technologies (SMARTapps) using Fast Health Interoperability Resource (FHIR) standard allow for open sharing and use of innovations across EHR systems. The aim of this project is to design and evaluate a SMARTapp on FHIR used across two large academic medical centers that exposes to physicians and nurses our new predictive data source from nursing documentation to increase care team situational awareness of at risk patients to decrease preventable adverse outcomes.

Communicating Narrative Concerns Entered by RNs (CONCERN) Clinical Decision Support (CDS) system is the application being designed and evaluated. CONCERN Intervention Trial Design will be a multiple time-series intervention. Baseline data will be collected at all study sites. Silent release mode (no SMARTapp notification) will be used in non-equivalent control units and as a post-intervention unit control to evaluate if notifying clinicians can decrease rates of length of stay on non-ICU units and rates of 30-day hospital readmissions. Different versions of the CDS system (SMARTapp) will be incorporated for dynamic, adaptive functionality and determine if the pattern of nursing documentation has changed. A "burn-in" phase is built in to evaluate adoption and adaptation to the algorithm and phases for deployment of the silent release mode within the multiple time-series intervention trial for a total of 18 months of data collection, including pre-intervention data collection and silent release modes.

ELIGIBILITY:
Study inclusion criteria for patients:

* Inpatients with a stay of at least 24 hours on one of our study units

Study exclusion criteria for patients:

* Inpatients with less than 24 hours on one of our study units
* Patients less than 18 years of age
* Hospice patients
* Did not have a hospital encounter, patients not on one of our study units.

Definition of Study Units:

A clinical unit is considered a CONCERN Study unit if it meets the following criteria:

* A general medical or surgical acute care or critical care unit

The following clinical units are NOT considered CONCERN Study units:

* Pediatric or Neonatal units
* Hospice units
* Emergency Department
* Oncology units
* Obstetrician (OB)/labor and delivery units
* Behavioral/psych units
* Observational units
* Operating room
* Pre-op
* Post-op/Post Anesthesia Care Unit (PACU)
* Same day surgical units
* Plastics units
* Virtual departments in EHR database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60893 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Dykes, PhD, Principal Investigator — Brigham and Women's Hospital; Sarah Collins Rossetti, PhD, Principal Investigator — Columbia University; Kenrick Cato, PhD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - New York Presbyterian Columbia University Medical Center, New York, New York
  - New York Presbyterian Allen Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No
This study will develop an open source SmartApp using interoperability standards. The investigators will make all source code available to any researchers upon request. This approach will ensure open access to all project aims, methods, resources, and deliverables by anyone via a study web-page. To aid in replication this web-page will include methods as well as other project processes such as stakeholder engagement, technical development, governance and lessons learned.

REFERENCES:
- [Background] Hripcsak G, Zhou L, Parsons S, Das AK, Johnson SB. Modeling electronic discharge summaries as a simple temporal constraint satisfaction problem. J Am Med Inform Assoc. 2005 Jan-Feb;12(1):55-63. doi: 10.1197/jamia.M1623. Epub 2004 Oct 18. PMID 15492038
- [Background] Zhou L, Parsons S, Hripcsak G. The evaluation of a temporal reasoning system in processing clinical discharge summaries. J Am Med Inform Assoc. 2008 Jan-Feb;15(1):99-106. doi: 10.1197/jamia.M2467. Epub 2007 Oct 18. PMID 17947618
- [Background] Sittig DF, Wright A, Osheroff JA, Middleton B, Teich JM, Ash JS, Campbell E, Bates DW. Grand challenges in clinical decision support. J Biomed Inform. 2008 Apr;41(2):387-92. doi: 10.1016/j.jbi.2007.09.003. Epub 2007 Sep 21. PMID 18029232
- [Background] Hripcsak G, Elhadad N, Chen YH, Zhou L, Morrison FP. Using empiric semantic correlation to interpret temporal assertions in clinical texts. J Am Med Inform Assoc. 2009 Mar-Apr;16(2):220-7. doi: 10.1197/jamia.M3007. Epub 2008 Dec 11. PMID 19074297
- [Background] Muller-Engelmann M, Krones T, Keller H, Donner-Banzhoff N. Decision making preferences in the medical encounter--a factorial survey design. BMC Health Serv Res. 2008 Dec 17;8:260. doi: 10.1186/1472-6963-8-260. PMID 19091091
- [Background] Murphy SN, Weber G, Mendis M, Gainer V, Chueh HC, Churchill S, Kohane I. Serving the enterprise and beyond with informatics for integrating biology and the bedside (i2b2). J Am Med Inform Assoc. 2010 Mar-Apr;17(2):124-30. doi: 10.1136/jamia.2009.000893. PMID 20190053
- [Background] Albers DJ, Hripcsak G. A statistical dynamics approach to the study of human health data: resolving population scale diurnal variation in laboratory data. Phys Lett A. 2010 Feb 15;374(9):1159-1164. doi: 10.1016/j.physleta.2009.12.067. PMID 20544004
- [Background] Collins SA, Bakken S, Vawdrey DK, Coiera E, Currie L. Model development for EHR interdisciplinary information exchange of ICU common goals. Int J Med Inform. 2011 Aug;80(8):e141-9. doi: 10.1016/j.ijmedinf.2010.09.009. Epub 2010 Oct 25. PMID 20974549
- [Background] Collins SA, Bakken S, Vawdrey DK, Coiera E, Currie LM. Agreement between common goals discussed and documented in the ICU. J Am Med Inform Assoc. 2011 Jan-Feb;18(1):45-50. doi: 10.1136/jamia.2010.006437. Epub 2010 Nov 27. PMID 21113075
- [Background] Hripcsak G, Vawdrey DK, Fred MR, Bostwick SB. Use of electronic clinical documentation: time spent and team interactions. J Am Med Inform Assoc. 2011 Mar-Apr;18(2):112-7. doi: 10.1136/jamia.2010.008441. Epub 2011 Feb 2. PMID 21292706
- [Background] Senathirajah Y, Bakken S. Visual clustering analysis of CIS logs to inform creation of a user-configurable Web CIS interface. Methods Inf Med. 2011;50(4):337-48. doi: 10.3414/ME09-01-0087. Epub 2011 Jun 21. PMID 21691676
- [Background] Merchant RM, Yang L, Becker LB, Berg RA, Nadkarni V, Nichol G, Carr BG, Mitra N, Bradley SM, Abella BS, Groeneveld PW; American Heart Association Get With The Guidelines-Resuscitation Investigators. Incidence of treated cardiac arrest in hospitalized patients in the United States. Crit Care Med. 2011 Nov;39(11):2401-6. doi: 10.1097/CCM.0b013e3182257459. PMID 21705896
- [Background] Collins SA, Vawdrey DK. "Reading between the lines" of flow sheet data: nurses' optional documentation associated with cardiac arrest outcomes. Appl Nurs Res. 2012 Nov;25(4):251-7. doi: 10.1016/j.apnr.2011.06.002. Epub 2011 Nov 12. PMID 22079746
- [Background] Hripcsak G, Albers DJ, Perotte A. Exploiting time in electronic health record correlations. J Am Med Inform Assoc. 2011 Dec;18 Suppl 1(Suppl 1):i109-15. doi: 10.1136/amiajnl-2011-000463. Epub 2011 Nov 23. PMID 22116643
- [Background] Mandl KD, Mandel JC, Murphy SN, Bernstam EV, Ramoni RL, Kreda DA, McCoy JM, Adida B, Kohane IS. The SMART Platform: early experience enabling substitutable applications for electronic health records. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):597-603. doi: 10.1136/amiajnl-2011-000622. Epub 2012 Mar 17. PMID 22427539
- [Background] Vawdrey DK, Wilcox LG, Collins S, Feiner S, Mamykina O, Stein DM, Bakken S, Fred MR, Stetson PD. Awareness of the Care Team in Electronic Health Records. Appl Clin Inform. 2011;2(4):395-405. doi: 10.4338/ACI-2011-05-RA-0034. PMID 22574103
- [Background] Rothman MJ, Solinger AB, Rothman SI, Finlay GD. Clinical implications and validity of nursing assessments: a longitudinal measure of patient condition from analysis of the Electronic Medical Record. BMJ Open. 2012 Aug 8;2(4):e000646. doi: 10.1136/bmjopen-2012-000849. Print 2012. PMID 22874626
- [Background] Zhou L, Karipineni N, Lewis J, Maviglia SM, Fairbanks A, Hongsermeier T, Middleton B, Rocha RA. A study of diverse clinical decision support rule authoring environments and requirements for integration. BMC Med Inform Decis Mak. 2012 Nov 12;12:128. doi: 10.1186/1472-6947-12-128. PMID 23145874
- [Background] Brady PW, Muething S, Kotagal U, Ashby M, Gallagher R, Hall D, Goodfriend M, White C, Bracke TM, DeCastro V, Geiser M, Simon J, Tucker KM, Olivea J, Conway PH, Wheeler DS. Improving situation awareness to reduce unrecognized clinical deterioration and serious safety events. Pediatrics. 2013 Jan;131(1):e298-308. doi: 10.1542/peds.2012-1364. Epub 2012 Dec 10. PMID 23230078
- [Background] Albers DJ, Hripcsak G, Schmidt M. Population physiology: leveraging electronic health record data to understand human endocrine dynamics. PLoS One. 2012;7(12):e48058. doi: 10.1371/journal.pone.0048058. Epub 2012 Dec 14. PMID 23272040
- [Background] Fukui S, Salyers MP, Matthias MS, Collins L, Thompson J, Coffman M, Torrey WC. Predictors of shared decision making and level of agreement between consumers and providers in psychiatric care. Community Ment Health J. 2014 May;50(4):375-82. doi: 10.1007/s10597-012-9584-0. Epub 2013 Jan 9. PMID 23299226
- [Background] Middleton B, Bloomrosen M, Dente MA, Hashmat B, Koppel R, Overhage JM, Payne TH, Rosenbloom ST, Weaver C, Zhang J; American Medical Informatics Association. Enhancing patient safety and quality of care by improving the usability of electronic health record systems: recommendations from AMIA. J Am Med Inform Assoc. 2013 Jun;20(e1):e2-8. doi: 10.1136/amiajnl-2012-001458. Epub 2013 Jan 25. PMID 23355463
- [Background] Smith SW, Koppel R. Healthcare information technology's relativity problems: a typology of how patients' physical reality, clinicians' mental models, and healthcare information technology differ. J Am Med Inform Assoc. 2014 Jan-Feb;21(1):117-31. doi: 10.1136/amiajnl-2012-001419. Epub 2013 Jun 25. PMID 23800960
- [Background] Finlay GD, Rothman MJ, Smith RA. Measuring the modified early warning score and the Rothman index: advantages of utilizing the electronic medical record in an early warning system. J Hosp Med. 2014 Feb;9(2):116-9. doi: 10.1002/jhm.2132. Epub 2013 Dec 19. PMID 24357519
- [Background] Cato K, Hyun S, Bakken S. Response to a mobile health decision-support system for screening and management of tobacco use. Oncol Nurs Forum. 2014 Mar 1;41(2):145-52. doi: 10.1188/14.ONF.145-152. PMID 24578074
- [Background] Mandl KD, Kohane IS, McFadden D, Weber GM, Natter M, Mandel J, Schneeweiss S, Weiler S, Klann JG, Bickel J, Adams WG, Ge Y, Zhou X, Perkins J, Marsolo K, Bernstam E, Showalter J, Quarshie A, Ofili E, Hripcsak G, Murphy SN. Scalable Collaborative Infrastructure for a Learning Healthcare System (SCILHS): architecture. J Am Med Inform Assoc. 2014 Jul-Aug;21(4):615-20. doi: 10.1136/amiajnl-2014-002727. Epub 2014 May 12. PMID 24821734
- [Background] Albers DJ, Elhadad N, Tabak E, Perotte A, Hripcsak G. Dynamical phenotyping: using temporal analysis of clinically collected physiologic data to stratify populations. PLoS One. 2014 Jun 16;9(6):e96443. doi: 10.1371/journal.pone.0096443. eCollection 2014. PMID 24933368
- [Background] Zhou L, Lu Y, Vitale CJ, Mar PL, Chang F, Dhopeshwarkar N, Rocha RA. Representation of information about family relatives as structured data in electronic health records. Appl Clin Inform. 2014 Apr 9;5(2):349-67. doi: 10.4338/ACI-2013-10-RA-0080. eCollection 2014. PMID 25024754
- [Background] Hum RS, Cato K, Sheehan B, Patel S, Duchon J, DeLaMora P, Ferng YH, Graham P, Vawdrey DK, Perlman J, Larson E, Saiman L. Developing clinical decision support within a commercial electronic health record system to improve antimicrobial prescribing in the neonatal ICU. Appl Clin Inform. 2014 Apr 9;5(2):368-87. doi: 10.4338/ACI-2013-09-RA-0069. eCollection 2014. PMID 25024755
- [Background] Senathirajah Y, Bakken S, Kaufman D. The clinician in the Driver's Seat: part 1 - a drag/drop user-composable electronic health record platform. J Biomed Inform. 2014 Dec;52:165-76. doi: 10.1016/j.jbi.2014.09.002. Epub 2014 Sep 18. PMID 25240253
- [Background] Yakusheva O, Lindrooth R, Weiss M. Nurse value-added and patient outcomes in acute care. Health Serv Res. 2014 Dec;49(6):1767-86. doi: 10.1111/1475-6773.12236. Epub 2014 Sep 25. PMID 25256089
- [Background] Drew BJ, Harris P, Zegre-Hemsey JK, Mammone T, Schindler D, Salas-Boni R, Bai Y, Tinoco A, Ding Q, Hu X. Insights into the problem of alarm fatigue with physiologic monitor devices: a comprehensive observational study of consecutive intensive care unit patients. PLoS One. 2014 Oct 22;9(10):e110274. doi: 10.1371/journal.pone.0110274. eCollection 2014. PMID 25338067
- [Background] Klann JG, Mendis M, Phillips LC, Goodson AP, Rocha BH, Goldberg HS, Wattanasin N, Murphy SN. Taking advantage of continuity of care documents to populate a research repository. J Am Med Inform Assoc. 2015 Mar;22(2):370-9. doi: 10.1136/amiajnl-2014-003040. Epub 2014 Oct 28. PMID 25352566
- [Background] Senathirajah Y, Kaufman D, Bakken S. The clinician in the driver's seat: part 2 - intelligent uses of space in a drag/drop user-composable electronic health record. J Biomed Inform. 2014 Dec;52:177-88. doi: 10.1016/j.jbi.2014.09.008. Epub 2014 Oct 24. PMID 25445921
- [Background] Hripcsak G, Albers DJ, Perotte A. Parameterizing time in electronic health record studies. J Am Med Inform Assoc. 2015 Jul;22(4):794-804. doi: 10.1093/jamia/ocu051. Epub 2015 Feb 26. PMID 25725004
- [Background] Adler L, Yi D, Li M, McBroom B, Hauck L, Sammer C, Jones C, Shaw T, Classen D. Impact of Inpatient Harms on Hospital Finances and Patient Clinical Outcomes. J Patient Saf. 2018 Jun;14(2):67-73. doi: 10.1097/PTS.0000000000000171. PMID 25803176
- [Background] Payne TH, Corley S, Cullen TA, Gandhi TK, Harrington L, Kuperman GJ, Mattison JE, McCallie DP, McDonald CJ, Tang PC, Tierney WM, Weaver C, Weir CR, Zaroukian MH. Report of the AMIA EHR-2020 Task Force on the status and future direction of EHRs. J Am Med Inform Assoc. 2015 Sep;22(5):1102-10. doi: 10.1093/jamia/ocv066. Epub 2015 May 28. No abstract available. PMID 26024883
- [Background] Cato KD, Cohen B, Larson E. Data elements and validation methods used for electronic surveillance of health care-associated infections: a systematic review. Am J Infect Control. 2015 Jun;43(6):600-5. doi: 10.1016/j.ajic.2015.02.006. PMID 26042848
- [Background] Schulz CM, Krautheim V, Hackemann A, Kreuzer M, Kochs EF, Wagner KJ. Situation awareness errors in anesthesia and critical care in 200 cases of a critical incident reporting system. BMC Anesthesiol. 2016 Jan 16;16:4. doi: 10.1186/s12871-016-0172-7. PMID 26772179
- [Background] Liu V, Escobar GJ, Greene JD, Soule J, Whippy A, Angus DC, Iwashyna TJ. Hospital deaths in patients with sepsis from 2 independent cohorts. JAMA. 2014 Jul 2;312(1):90-2. doi: 10.1001/jama.2014.5804. No abstract available. PMID 24838355
- [Background] Sharek PJ, Parast LM, Leong K, Coombs J, Earnest K, Sullivan J, Frankel LR, Roth SJ. Effect of a rapid response team on hospital-wide mortality and code rates outside the ICU in a Children's Hospital. JAMA. 2007 Nov 21;298(19):2267-74. doi: 10.1001/jama.298.19.2267. PMID 18029830
- [Background] Hiissa M, Pahikkala T, Suominen H, Lehtikunnas T, Back B, Karsten H, Salantera S, Salakoski T. Towards automated classification of intensive care nursing narratives. Int J Med Inform. 2007 Dec;76 Suppl 3:S362-8. doi: 10.1016/j.ijmedinf.2007.03.003. Epub 2007 May 21. PMID 17513166
- [Background] Goodwin L, VanDyne M, Lin S, Talbert S. Data mining issues and opportunities for building nursing knowledge. J Biomed Inform. 2003 Aug-Oct;36(4-5):379-88. doi: 10.1016/j.jbi.2003.09.020. PMID 14643734
- [Background] Zhou L, Hripcsak G. Temporal reasoning with medical data--a review with emphasis on medical natural language processing. J Biomed Inform. 2007 Apr;40(2):183-202. doi: 10.1016/j.jbi.2006.12.009. Epub 2007 Jan 11. PMID 17317332
- [Background] Hazlehurst B, McMullen CK, Gorman PN. Distributed cognition in the heart room: how situation awareness arises from coordinated communications during cardiac surgery. J Biomed Inform. 2007 Oct;40(5):539-51. doi: 10.1016/j.jbi.2007.02.001. Epub 2007 Feb 8. PMID 17368112
- [Background] Zhou L, Plasek JM, Mahoney LM, Chang FY, DiMaggio D, Rocha RA. Mapping Partners Master Drug Dictionary to RxNorm using an NLP-based approach. J Biomed Inform. 2012 Aug;45(4):626-33. doi: 10.1016/j.jbi.2011.11.006. Epub 2011 Nov 28. PMID 22142948
- [Background] Lai KH, Topaz M, Goss FR, Zhou L. Automated misspelling detection and correction in clinical free-text records. J Biomed Inform. 2015 Jun;55:188-95. doi: 10.1016/j.jbi.2015.04.008. Epub 2015 Apr 24. PMID 25917057
- [Background] McNeill G, Bryden D. Do either early warning systems or emergency response teams improve hospital patient survival? A systematic review. Resuscitation. 2013 Dec;84(12):1652-67. doi: 10.1016/j.resuscitation.2013.08.006. Epub 2013 Aug 17. PMID 23962485
- [Background] Alam N, Hobbelink EL, van Tienhoven AJ, van de Ven PM, Jansma EP, Nanayakkara PW. The impact of the use of the Early Warning Score (EWS) on patient outcomes: a systematic review. Resuscitation. 2014 May;85(5):587-94. doi: 10.1016/j.resuscitation.2014.01.013. Epub 2014 Jan 25. PMID 24467882
- [Background] Wahl WL, Talsma A, Dawson C, Dickinson S, Pennington K, Wilson D, Arbabi S, Taheri PA. Use of computerized ICU documentation to capture ICU core measures. Surgery. 2006 Oct;140(4):684-9; discussion 690. doi: 10.1016/j.surg.2006.06.017. Epub 2006 Sep 6. PMID 17011917
- [Background] Rittenhouse DR, Shortell SM, Fisher ES. Primary care and accountable care--two essential elements of delivery-system reform. N Engl J Med. 2009 Dec 10;361(24):2301-3. doi: 10.1056/NEJMp0909327. No abstract available. PMID 19864649
- [Background] Berwick DM. Launching accountable care organizations--the proposed rule for the Medicare Shared Savings Program. N Engl J Med. 2011 Apr 21;364(16):e32. doi: 10.1056/NEJMp1103602. Epub 2011 Mar 31. No abstract available. PMID 21452999
- [Background] Cioffi J. Recognition of patients who require emergency assistance: a descriptive study. Heart Lung. 2000 Jul-Aug;29(4):262-8. doi: 10.1067/mhl.2000.108327. PMID 10900063
- [Background] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Background] Alterovitz G, Warner J, Zhang P, Chen Y, Ullman-Cullere M, Kreda D, Kohane IS. SMART on FHIR Genomics: facilitating standardized clinico-genomic apps. J Am Med Inform Assoc. 2015 Nov;22(6):1173-8. doi: 10.1093/jamia/ocv045. Epub 2015 Jul 21. PMID 26198304
- [Background] Devita MA, Bellomo R, Hillman K, Kellum J, Rotondi A, Teres D, Auerbach A, Chen WJ, Duncan K, Kenward G, Bell M, Buist M, Chen J, Bion J, Kirby A, Lighthall G, Ovreveit J, Braithwaite RS, Gosbee J, Milbrandt E, Peberdy M, Savitz L, Young L, Harvey M, Galhotra S. Findings of the first consensus conference on medical emergency teams. Crit Care Med. 2006 Sep;34(9):2463-78. doi: 10.1097/01.CCM.0000235743.38172.6E. PMID 16878033
- [Background] Schulz CM, Endsley MR, Kochs EF, Gelb AW, Wagner KJ. Situation awareness in anesthesia: concept and research. Anesthesiology. 2013 Mar;118(3):729-42. doi: 10.1097/ALN.0b013e318280a40f. PMID 23291626
- [Background] Matney S, Brewster PJ, Sward KA, Cloyes KG, Staggers N. Philosophical approaches to the nursing informatics data-information-knowledge-wisdom framework. ANS Adv Nurs Sci. 2011 Jan-Mar;34(1):6-18. doi: 10.1097/ANS.0b013e3182071813. PMID 21150551
- [Background] Hermanides J, Vriesendorp TM, Bosman RJ, Zandstra DF, Hoekstra JB, Devries JH. Glucose variability is associated with intensive care unit mortality. Crit Care Med. 2010 Mar;38(3):838-42. doi: 10.1097/CCM.0b013e3181cc4be9. PMID 20035218
- [Background] Egi M, Bellomo R, Stachowski E, French CJ, Hart GK, Taori G, Hegarty C, Bailey M. The interaction of chronic and acute glycemia with mortality in critically ill patients with diabetes. Crit Care Med. 2011 Jan;39(1):105-11. doi: 10.1097/CCM.0b013e3181feb5ea. PMID 20975552
- [Background] Watson A, Skipper C, Steury R, Walsh H, Levin A. Inpatient nursing care and early warning scores: a workflow mismatch. J Nurs Care Qual. 2014 Jul-Sep;29(3):215-22. doi: 10.1097/NCQ.0000000000000058. PMID 24569518
- [Background] James JT. A new, evidence-based estimate of patient harms associated with hospital care. J Patient Saf. 2013 Sep;9(3):122-8. doi: 10.1097/PTS.0b013e3182948a69. PMID 23860193
- [Background] Albers DJ, Sprott JC, Crutchfield JP. Persistent chaos in high dimensions. Phys Rev E Stat Nonlin Soft Matter Phys. 2006 Nov;74(5 Pt 2):057201. doi: 10.1103/PhysRevE.74.057201. Epub 2006 Nov 2. PMID 17280024
- [Background] Nakamura A, Osonoi T, Terauchi Y. Relationship between urinary sodium excretion and pioglitazone-induced edema. J Diabetes Investig. 2010 Oct 19;1(5):208-11. doi: 10.1111/j.2040-1124.2010.00046.x. PMID 24843434
- [Background] Jones L, King L, Wilson C. A literature review: factors that impact on nurses' effective use of the Medical Emergency Team (MET). J Clin Nurs. 2009 Dec;18(24):3379-90. doi: 10.1111/j.1365-2702.2009.02944.x. PMID 20487489
- [Background] Bates DW, Saria S, Ohno-Machado L, Shah A, Escobar G. Big data in health care: using analytics to identify and manage high-risk and high-cost patients. Health Aff (Millwood). 2014 Jul;33(7):1123-31. doi: 10.1377/hlthaff.2014.0041. PMID 25006137
- [Background] Churpek MM, Yuen TC, Park SY, Gibbons R, Edelson DP. Using electronic health record data to develop and validate a prediction model for adverse outcomes in the wards*. Crit Care Med. 2014 Apr;42(4):841-8. doi: 10.1097/CCM.0000000000000038. PMID 24247472
- [Background] Zhang AL, Chen RX, Kang MF, Fan HL, Wang WL. Study of the regulatory effect of acupuncture on rotation-induced gastric dysrhythmia in rabbits. World J Gastroenterol. 1997 Mar 15;3(1):54-5. doi: 10.3748/wjg.v3.i1.54. PMID 27006588
- [Background] Collins S, Bakken S, Vawdrey D, Coiera E, Currie LM. Discuss now, document later: CIS/CPOE perceived to be a 'shift behind' in the ICU. Stud Health Technol Inform. 2010;160(Pt 1):178-82. PMID 20841673
- [Background] Zhou L, Hongsermeier T, Boxwala A, Lewis J, Kawamoto K, Maviglia S, Gentile D, Teich JM, Rocha R, Bell D, Middleton B. Structured representation for core elements of common clinical decision support interventions to facilitate knowledge sharing. Stud Health Technol Inform. 2013;192:195-9. PMID 23920543
- [Background] Zhou L, Friedman C, Parsons S, Hripcsak G. System architecture for temporal information extraction, representation and reasoning in clinical narrative reports. AMIA Annu Symp Proc. 2005;2005:869-73. PMID 16779164
- [Background] Collins SA, Cato K, Albers D, Scott K, Stetson PD, Bakken S, Vawdrey DK. Relationship between nursing documentation and patients' mortality. Am J Crit Care. 2013 Jul;22(4):306-13. doi: 10.4037/ajcc2013426. PMID 23817819
- [Background] Collins SA, Fred M, Wilcox L, Vawdrey DK. Workarounds used by nurses to overcome design constraints of electronic health records. NI 2012 (2012). 2012 Jun 23;2012:93. eCollection 2012. PMID 24199061
- [Background] Collins SA, Currie LM. Interdisciplinary communication in the ICU. Stud Health Technol Inform. 2009;146:362-6. PMID 19592866
- [Background] Collins S, Hurley AC, Chang FY, Illa AR, Benoit A, Laperle S, Dykes PC. Content and functional specifications for a standards-based multidisciplinary rounding tool to maintain continuity across acute and critical care. J Am Med Inform Assoc. 2014 May-Jun;21(3):438-47. doi: 10.1136/amiajnl-2013-001949. Epub 2013 Sep 30. PMID 24081019
- [Background] Collins SA, Gazarian P, Stade D, McNally K, Morrison C, Ohashi K, Lehmann L, Dalal A, Bates DW, Dykes PC. Clinical Workflow Observations to Identify Opportunities for Nurse, Physicians and Patients to Share a Patient-centered Plan of Care. AMIA Annu Symp Proc. 2014 Nov 14;2014:414-23. eCollection 2014. PMID 25954345
- [Background] Ferguson TB Jr. The Institute of Medicine committee report "best care at lower cost: the path to continuously learning health care". Circ Cardiovasc Qual Outcomes. 2012 Nov;5(6):e93-4. doi: 10.1161/CIRCOUTCOMES.112.968768. No abstract available. PMID 23170008
- [Background] Albers DJ, Hripcsak G. Using time-delayed mutual information to discover and interpret temporal correlation structure in complex populations. Chaos. 2012 Mar;22(1):013111. doi: 10.1063/1.3675621. PMID 22462987
- [Background] Hyun S, Bakken S. Toward the creation of an ontology for nursing document sections: mapping section names to the LOINC semantic model. AMIA Annu Symp Proc. 2006;2006:364-8. PMID 17238364
- [Background] Aiken LH, Clarke SP, Sloane DM. Hospital staffing, organization, and quality of care: Cross-national findings. Nurs Outlook. 2002 Sep-Oct;50(5):187-94. doi: 10.1067/mno.2002.126696. PMID 12386653
- [Background] Moss J, Andison M, Sobko H. An analysis of narrative nursing documentation in an otherwise structured intensive care clinical information system. AMIA Annu Symp Proc. 2007 Oct 11;2007:543-7. PMID 18693895
- [Background] Bequette BW. Algorithms for a closed-loop artificial pancreas: the case for model predictive control. J Diabetes Sci Technol. 2013 Nov 1;7(6):1632-43. doi: 10.1177/193229681300700624. PMID 24351190
- [Background] Zhou L, Plasek JM, Mahoney LM, Karipineni N, Chang F, Yan X, Chang F, Dimaggio D, Goldman DS, Rocha RA. Using Medical Text Extraction, Reasoning and Mapping System (MTERMS) to process medication information in outpatient clinical notes. AMIA Annu Symp Proc. 2011;2011:1639-48. Epub 2011 Oct 22. PMID 22195230
- [Background] Stein-Parbury J, Liaschenko J. Understanding collaboration between nurses and physicians as knowledge at work. Am J Crit Care. 2007 Sep;16(5):470-7; quiz 478. PMID 17724244
- [Background] Collins S, Bakken S, Cimino JJ, Currie LM. Identifying logical clinical context clusters in nursing orders for the purpose of information retrieval. AMIA Annu Symp Proc. 2008 Nov 6;2008:131-5. PMID 18999260
- [Background] Senathirajah Y, Kaufman D, Bakken S. Essential questions: accuracy, errors and user perceptions in a drag/drop user-composable electronic health record. Stud Health Technol Inform. 2013;194:181-7. PMID 23941953
- [Background] Currie L, Sheehan B, Graham PL 3rd, Stetson P, Cato K, Wilcox A. Sociotechnical analysis of a neonatal ICU. Stud Health Technol Inform. 2009;146:258-62. PMID 19592845
- [Background] Cato KD, Bakken S. What am I giving tonight? Information needs of nurses related to patient medications administration while using a clinical information system. NI 2012 (2012). 2012 Jun 23;2012:65. eCollection 2012. PMID 24199053
- [Background] Topaz M, Seger DL, Lai K, Wickner PG, Goss F, Dhopeshwarkar N, Chang F, Bates DW, Zhou L. High Override Rate for Opioid Drug-allergy Interaction Alerts: Current Trends and Recommendations for Future. Stud Health Technol Inform. 2015;216:242-6. PMID 26262047
- [Background] Klann JG, Phillips LC, Herrick C, Joss MAH, Wagholikar KB, Murphy SN. Web services for data warehouses: OMOP and PCORnet on i2b2. J Am Med Inform Assoc. 2018 Oct 1;25(10):1331-1338. doi: 10.1093/jamia/ocy093. PMID 30085008
- [Background] Sedigh-Sarvestani M, Albers DJ, Gluckman BJ. Data assimilation of glucose dynamics for use in the intensive care unit. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:5437-40. doi: 10.1109/EMBC.2012.6347224. PMID 23367159
- [Background] Ludwick R, Zeller RA. The factorial survey: an experimental method to replicate real world problems. Nurs Res. 2001 Mar-Apr;50(2):129-33. doi: 10.1097/00006199-200103000-00009. PMID 11302293
- [Derived] Rossetti SC, Dykes PC, Knaplund C, Cho S, Withall J, Lowenthal G, Albers D, Lee RY, Jia H, Bakken S, Kang MJ, Chang FY, Zhou L, Bates DW, Daramola T, Liu F, Schwartz-Dillard J, Tran M, Bokhari SMA, Thate J, Cato KD. Real-time surveillance system for patient deterioration: a pragmatic cluster-randomized controlled trial. Nat Med. 2025 Jun;31(6):1895-1902. doi: 10.1038/s41591-025-03609-7. Epub 2025 Apr 2. PMID 40175738
- [Derived] Rossetti SC, Dykes PC, Knaplund C, Cho S, Withall J, Lowenthal G, Albers D, Lee R, Jia H, Bakken S, Kang MJ, Chang FY, Zhou L, Bates DW, Daramola T, Liu F, Schwartz-Dillard J, Tran M, Abbas Bokhari SM, Thate J, Cato KD. Multisite Pragmatic Cluster-Randomized Controlled Trial of the CONCERN Early Warning System. medRxiv [Preprint]. 2024 Jun 4:2024.06.04.24308436. doi: 10.1101/2024.06.04.24308436. PMID 38883706
- [Derived] Rossetti SC, Dykes PC, Knaplund C, Kang MJ, Schnock K, Garcia JP Jr, Fu LH, Chang F, Thai T, Fred M, Korach TZ, Zhou L, Klann JG, Albers D, Schwartz J, Lowenthal G, Jia H, Liu F, Cato K. The Communicating Narrative Concerns Entered by Registered Nurses (CONCERN) Clinical Decision Support Early Warning System: Protocol for a Cluster Randomized Pragmatic Clinical Trial. JMIR Res Protoc. 2021 Dec 10;10(12):e30238. doi: 10.2196/30238. PMID 34889766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Clusters were the individual clinical units across the four hospitals that included all non-specialty acute care units (ACUs) and intensive care units (ICUs).
Units Other Than Participants: clinical unit
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 27869; 37 clinical unit | 33024; 37 clinical unit
Completed | 27869; 37 clinical unit | 33024; 37 clinical unit
Not Completed | 0; 0 clinical unit | 0; 0 clinical unit

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 27,869 | 33,024 | 60893
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.67 (17.10) | 62.62 (17.56) | 63.1 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13,903 | 16,968 | 30871
  Male | 13,966 | 16,056 | 30022
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5,903 | 7,442 | 13345
  Not Hispanic or Latino | 20,304 | 23,618 | 43922
  Unknown or Not Reported | 1,662 | 1,964 | 3626
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 634 | 703 | 1337
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4,224 | 4,878 | 9102
  White | 16,278 | 18,923 | 35201
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6,733 | 8,520 | 15253
Region of Enrollment [Number; unit: participants]
  United States | 27,869 | 33,024 | 60893
Primary language English [Count of Participants; unit: Participants] | 22,584 | 26,713 | 49297
Clinical unit type [Count of Participants; unit: Participants]
  ACU | 25,704 | 31,050 | 56754
  ICU | 2,165 | 1,974 | 4139

OUTCOME MEASURES:

1. Primary Outcome: In-hospital Mortalities
Description: Number of patient deaths occurring in the hospital.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- CONCERN Intervention Group: Experimental data will be collected in the CONCERN CDS system that will be "live" in the EHR in "active" release mode (e.g., providing CONCERN CDS system notification to clinicians).
- Usual Care Group: Control data will be collected in the CONCERN CDS system that will be "live" in the EHR, but in silent release mode (e.g., not providing notification to clinicians).
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
Participants | 181 | 265

2. Primary Outcome: Average Length of Hospital Stay
Description: The number of days that a patient was in the hospital
Time Frame: Up to 24 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
days | 6.6 (0.82) | 7.2 (0.9)

3. Secondary Outcome: Number of Cardiac Arrests
Description: Cardiopulmonary events during hospitalization
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
Participants | 123 | 128

4. Secondary Outcome: Number of Hospital Acquired Sepsis
Description: Sepsis occurring during hospitalization
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
Participants | 1,461 | 1,578

5. Secondary Outcome: Number of Unanticipated Transfers to ICU
Description: Transfer to ICU from acute care study units during hospitalization
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
Participants | 505 | 377

6. Secondary Outcome: Number of Hospital Readmissions
Description: Readmission to the hospital within 30 days of being discharged alive.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | CONCERN Intervention Group | Usual Care Group
Number analyzed (Participants) | 33,024 | 27,869
Participants | 2,544 | 2,234

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | CONCERN Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 181/33024 | 265/27869
Serious Adverse Events (participants affected / at risk) | 0/33024 | 0/27869
Other Adverse Events (participants affected / at risk) | 0/33024 | 0/27869

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03911687/Prot_SAP_000.pdf